CLINICAL TRIAL: NCT05134012
Title: A Phase 3, Multicenter, Open Label Study to Confirm the Diagnostic Potential of Intravenously Administered [15-O]-H2O to Identify Coronary Artery Disease During Pharmacological Stress and Resting Conditions Using PET Imaging (RAPID-WATER-FLOW)
Brief Title: RAdiolabeled Perfusion to Identify Coronary Artery Disease Using WAter To Evaluate Responses of Myocardial FLOW (RAPID-WATER-FLOW)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MedTrace Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MedTrace-002
Record Dates: First submitted 2021-10-29; First posted 2021-11-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease
Keywords: Myocardial Blood Flow (MBF); Myocardial Perfusion Imaging (MPI); RAPID-WATER-FLOW; Positron Emission Tomography (PET); Oxygen-15; Coronary Artery Disease (CAD)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Approximately 182 evaluable participants with suspected CAD referred for testing will be included in the study. All participants will receive two doses of [15-O]-H2O as part of a single PET imaging session (one dose at rest and one during pharmacological stress with adenosine).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- [O-15]-Water PET Myocardial Perfusion Imaging (MPI) (Experimental): All participants with suspected CAD will receive two doses of [15-O]-H2O as part of a single PET imaging session (one dose at rest and one during pharmacological stress with adenosine).
  Interventions: Drug: [O-15]-Water PET Myocardial Perfusion Imaging (MPI)

INTERVENTIONS:
Drug: [O-15]-Water PET Myocardial Perfusion Imaging (MPI) — [15-O]-H2O injection is a novel PET imaging agent labeled with the radioisotope [15-O] administered as an intravenous (IV) injection. Participants will receive [15-O]-H2O treatment twice as a part of a single day imaging session. All participants will receive two IV boluses of [15-O]-H2O injection in a peripheral vein; one at rest and one during pharmacological stress.

SUMMARY:
This a Phase 3, prospective, open-label, multicenter study of [15-O]-H2O injection for PET imaging of subjects with suspected CAD. Approximately 182 evaluable participants with suspected CAD referred for testing will be included in the study at approximately 10 study sites in the United States and Europe. Approximately 215 participants will be enrolled to account for an estimated 15% drop-out rate. Screening assessments will occur prior to enrollment to confirm eligibility. All participants will receive two doses of [15-O]-H2O as part of a single PET imaging session (one dose at rest and one during pharmacological stress with adenosine). A safety follow-up phone call will occur 24 ± 8 hrs after completion of the [15-O]-H2O scan.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants ≥18 years;
2. Informed consent form (ICF) read, signed, and dated prior to any study procedures being performed;
3. Participants who fall into any one of the following categories:

   1. Have been referred for an ICA directly of after non-invasive testing (e.g., SPECT or PET MPI, stress echo, CCTA, ETT).
   2. Had an ICA with no intervention. However, if any stenosis >40% but ≤70% was observed, an FFR or iFR assessment was performed.
   3. Had a CCTA with normal coronaries or minimal CAD (no stenosis >25%).

   The SPECT study, PET 15O-H2O study, and ICA or CCTA testing need to be completed within a 30-day window, with time 0 defined as the date of the first of these three tests.
4. Women of Child Bearing Potential (WOCBP) must be non-pregnant, and non-lactating. For women of childbearing potential, the results of a urine human chorionic gonadotropin (HCG) pregnancy test (with the result known on the day of drug administration) must be negative; these participants must be practicing appropriate birth control from time of the screening visit until the end of the follow-up period. For women who are either surgically sterile (have a documented bilateral tubal ligation or oophorectomy and/or hysterectomy) or are post-menopausal (cessation of menses for more than 1 year), enrollment in the study without a pregnancy test at screening is allowed.
5. Male will need to use contraceptive methods until end of the follow-up period.
6. Participants are able to comply with all study procedures as described in the protocol.

Exclusion Criteria:

1. Participants are unable to undergo (even partially) any of the imaging procedures;
2. Participants with a known history of cardiac disease including:

   1. myocardial infarction, previous coronary revascularization, or chronic ischemic cardiomyopathy
   2. primary myocardial disease such as cardiac amyloidosis or hypertrophic cardiomyopathy
   3. known left ventricular dysfunction
   4. moderate or severe aortic or mitral stenosis or regurgitation
3. Participants in whom adenosine stress testing is contraindicated, including but not limited to:

   1. Participants with severe COPD or chronic asthma.
   2. Participants with second- or third-degree atrioventricular block without a pacemaker.
4. Participants with claustrophobia to an extent that would limit their ability to undergo SPECT and PET imaging (patients whose claustrophobia is known to be readily controlled with drugs or psychological support may be enrolled).
5. Participants who are on sildenafil (Viagra) or oral dipyridamole (Persantine, Aggrenox) therapy or on any PDE5 inhibitor (i.e. tadalafil, avanafil, vardenafil),and for whom its use cannot be terminated or suspended for ≥24 hours prior to treatment of study drug.
6. Participants with significant co-morbidities that would prevent appropriate completion of the protocol procedures.
7. Participants who have participated in another research study using investigational drugs within the 30 days prior to enrollment or through the duration of the trial (patients in observational studies with approved agents and participants known to be on placebo may be enrolled).
8. Participants who have previously participated in this study.
9. Subjects scheduled for, or planning to undergo, any interventional cardiac procedures between enrollment and ICA (pathway 1) or signing of informed consent and 15O-H2O PET MPI (pathway 2 and 3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Estimated)
Dates: Start 2022-05-08 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the [15-O]-H2O PET study using the truth-standard of ICA with FFR/iFR or CCTA. | 30 days
  Sensitivity and specificity are defined as follows:
  * True Positives (TP): Subjects with abnormal PET MPI and disease positive by the truth standard
  * True Negatives (TN): Subjects with normal PET MPI and disease negative by the truth standard
  * False Positives (FP): Subjects with abnormal PET MPI and disease negative by the truth standard
  * False Negatives (FN): Subjects with normal PET MPI and disease positive by the truth standard
  * Sensitivity: TP/(TP + FN)
  * Specificity: TN/(TN + FP)

SECONDARY OUTCOMES:
Sensitivity, specificity, and accuracy of [15-O]-H2O PET MPI in participants of special clinical interest (female, BMI≥30, diabetics, multivessel disease). | 30 days
  Sensitivity and specificity are defined as follows:
  * True Positives (TP): Subjects with abnormal PET MPI and disease positive by the truth standard
  * True Negatives (TN): Subjects with normal PET MPI and disease negative by the truth standard
  * False Positives (FP): Subjects with abnormal PET MPI and disease negative by the truth standard
  * False Negatives (FN): Subjects with normal PET MPI and disease positive by the truth standard
  * Sensitivity: TP/(TP + FN)
  * Specificity: TN/(TN + FP)
  * Accuracy: (TN + TP)/(TN + TP + FN + FP)
Adverse event analyses will include tabulations of the incidence (number and percent of subjects) with at least one TEAEs overall and by MedDRA system organ class (SOC) and preferred term (PT). This will be repeated for serious adverse. | 30 days
  Other Safety measures including the following will be summarized descriptively:
  1. ECG (ventricular heart rate, PR interval, QRS duration, QT interval, QTc interval)
  2. Vital Signs
  3. Concomitant Medications
  4. Protocol Deviations

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Borys, MD, Study Director — MedTrace Pharma A/S; Marcelo DiCarli, MD, Principal Investigator — Brigham and Women's Hospital
Locations (14):
- United States (7):
  - University of Iowa, Iowa City, Iowa
  - BAMF Healthcare, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada
- Aarhus University Hospital, Aarhus, Denmark
- Germany (2):
  - University Hospital Freiburg, Clinic for Nuclear Medicine, Freiburg im Breisgau
  - Department of Cardiology and Angiology -- Hannover Medical School (MHH), Hanover
- Amsterdam University Medical Center, Department of Radiology and Nuclear Medicine, Amsterdam, North Holland, Netherlands
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Norrland University Hospital Heart Center, Umeå

REFERENCES:
- [Derived] Di Carli MF, Gormsen LC, Chareonthaitawee P, Johnson GB, Beanlands R, DeKemp R, Schindler T, Gropler R, Kulkarni H, McNeely P, Soman P, Oz O, Zaha V, Sorensen J, Harms H, Orlandi C, Vandenbroucke E, Udelson J. Rationale and design of the RAPID-WATER-FLOW trial: Radiolabeled perfusion to identify coronary artery disease using water to evaluate responses of myocardial FLOW. J Nucl Cardiol. 2024 Jan;31:101779. doi: 10.1016/j.nuclcard.2023.101779. Epub 2023 Dec 5. PMID 38215598